CLINICAL TRIAL: NCT07216352
Title: Open-label Study Evaluating the Safety and Efficacy of AGE Serum in Non-menopausal Patients on Glucagon-like Peptide-1 Agonists
Brief Title: Evaluate the Safety and Efficacy of a Topical Serum (AGE Serum) in Improving Visible Signs of Aging
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Goldman, Butterwick, Fitzpatrick and Groff (Other)
Collaborators: L'Oreal (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGE-SERUM-2025
Record Dates: First submitted 2025-10-08; First posted 2025-10-14 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Laxity; Skin
Keywords: glp1; weight loss; skin laxity; skin texture; skin tone
MeSH Terms: conditions — Cutis Laxa; Weight Loss

STUDY DESIGN:
Intervention Model Description: All 25 adult subjects will be enrolled in to the same group and provided the same product.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AGE Product (Experimental): Enrolled subjects will received AGE Serum.
  Interventions: Other: AGE Serum

INTERVENTIONS:
Other: AGE Serum — AGE serum is a topical that contains a high concentration of 30% Proxylane and a synergistic blend of fruit-derived flavonoids (blueberry, pomegranate) and Cassia alata extract.

SUMMARY:
The primary objective is to evaluate the safety and efficacy of a topical serum (AGE serum) in improving visible signs of aging (e.g., fine lines, wrinkles, sagging, texture, radiance) on the full face and neck.The study will be conducted in non-menopausal female and male subjects who are on glucagon-like peptide-1 (GLP-1) agonist therapy for weight loss.

DETAILED DESCRIPTION:
enrolled subjects will apply a topical serum (AGE Serum) to the full face and neck twice daily for 12 weeks. Subject follow-up visits will occur at Week 6 and Week 12. Subjects will complete assessments and participate in and standardized 2D and 3D (Visia) digital photography.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of mild to moderate signs of facial aging (e.g., fine lines, laxity, dull texture) based on modified Griffith scale.
2. Adult men and women aged 25-50 years.
3. Fitzpatrick skin types I-IV.
4. Current treatment with a stable dose of GLP-1 agonist medication, including Ozempic, Rybelsus, or Wegovy for at least last 6 months.
5. Must be willing to sign a photography release and ICF, and complete the entire course of the study.
6. Subjects in good general health based on the investigator's judgment and medical history.
7. Negative urine pregnancy test result at the time of study entry (if applicable).
8. Subjects of childbearing potential must agree to use an effective method of birth control during the entire course of the study. All systemic birth control measures must be in consistent use for at least 30 days prior to study enrollment.

A. Acceptable forms of birth control are: oral contraceptive pill, injection, implant, patch, vaginal ring, intrauterine device/coil, double-barrier methods (e.g., sponge, spermicide, or condoms). Abstinence and/or vasectomized partners must agree to a second acceptable method of birth control (double-barrier) should the subject become sexually active.

B. A female is considered of non-childbearing potential if she is: postmenopausal (no menses for at least 12 months), without a uterus (hysterectomy) and/or both ovaries (oophorectomy), or bilateral tubal ligation.

Exclusion Criteria:

1. Pregnancy or planned pregnancy during the study or currently breastfeeding.
2. Current menopausal state.
3. Any uncontrolled systemic disease.
4. Current use of other GLP-1 agonist therapy aside from the GLP-1 agonist class of medications (Ozempic, Rybelsus, or Wegovy).
5. History of autoimmune connective tissue disease.
6. Current use of immunosuppressive medication.
7. Significant history or current evidence of a medical, psychological or other disorder that, in the investigator's opinion, would preclude enrollment into the study.
8. Active dermatitis or active infection in the proposed treatment area.
9. Mesotherapy; dermal fillers, biostimulator injectables; radiofrequency device treatments; microfocused ultrasound device treatments; laser and light-based device treatments; microneedling; cryolipolysis; high intensity focused electromagnetic energy device treatment; or surgery during the 12-month period before study treatment.
10. Creams/cosmeceuticals and/or home therapies for the prevention or treatment of skin quality in the treatment area during the 1-month period before study treatment.
11. Subjects with scarring in the treatment areas, which in the opinion of the investigator could impact results. Subjects with a history of keloids will be excluded.
12. Subjects who spray tanned or used sunless tanners in the treatment areas 1-month prior to study treatment.
13. History of bleeding disorder, concomitant use of anticoagulants, history of connective tissue disease (e.g., lupus, scleroderma), history of Bell's Palsy, epilepsy, smoking, and/or current pregnancy or breastfeeding.
14. Inability to ambulate following the procedure.
15. History of lidocaine and/or epinephrine sensitivity deemed by the investigator to preclude subject from enrolling into study.
16. Individuals with known allergies or sensitivities to any of the ingredients of any topical or injectable products being used in this study.
17. Current participation or participation within 30 days prior to the start of this study in a drug or other investigational research study.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-10-25 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Modified Griffith Scale | Baseline, Week 6 and Week12
  Modified Griffiths 10-point scale to be used for investigator grading of cutaneous signs of photoaging on the face.
  Global Fine Lines. Scale 0 (no fine lines) to 9 (numerous, many fine lines) Overall Hyperpigmentation: Scale 0 (no hyperpigmentation) to 9 (significant hyperpigmentation) Skin Tone Eveness: Scale 0 (very even tone) to 9 (uneven, discolored appearance) Skin Elasticity: Score 0 (skin feels toned and dense) to 9 (skin feels thin and flabby) Skin Firmness: Score 0 (firm, tight feeling) to 9 (loose, lax feeling) Skin Radiance: Score 0 (very radiant, luminous, glowing) to 9 (very dull) Skin Texture: Score 0 (very smooth) to 9 (very rough)

SECONDARY OUTCOMES:
Physician Global Aesthetic Improvement Scale | Week 12
  Physician Grading:
  1. Very Much Improved
  2. Much Improved
  3. Improved
  4. No Change
  5. Worse
Subject Global Aesthetic Improvement Scale | Week 12
  Subject Grading:
  1. Very Much Improved
  2. Much Improved
  3. Improved
  4. No Change
  5. Worse
Subject Self-Assessment Questionnaire | Baseline, Week 6 and Week 12
  Circle One
  Skin Feels More Comfortable:
  Agree Strongly Agree Neither Agree Disagree Disagree Disagree Strongly
  Skin Appears Younger Looking:
  Agree Strongly Agree Neither Agree Disagree Disagree Disagree Strongly
  Skin Appears Healthier:
  Agree Strongly Agree Neither Agree Disagree Disagree Disagree Strongly
  Skin Looks Renewed/Revitalized:
  Agree Strongly Agree Neither Agree Disagree Disagree Disagree Strongly
  Skin Looks Firmer:
  Agree Strongly Agree Neither Agree Disagree Disagree Disagree Strongly
  Skin Feels Elastic :
  Agree Strongly Agree Neither Agree Disagree Disagree Disagree Strongly
  Redness Looks Reduced:
  Agree Strongly Agree Neither Agree Disagree Disagree Disagree Strongly

CONTACTS AND LOCATIONS:
Locations (1):
- West Dermatology Research Center, San Diego, California, United States